CLINICAL TRIAL: NCT05609617
Title: Evaluation of Anti-aging Performance and Tolerance of a Hyaluronic Acid-based Filler NCTF135HA® Medical Device, on Filling the Superficial Wrinkles and on Skin Quality: HEBE2 Study
Brief Title: Evaluation of Anti-aging Performance and Tolerance of a Hyaluronic Acid-based Filler NCTF135HA®
Acronym: HEBE2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires FILLMED (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HEBE2: 2018-A03167-48; 2018-A03167-48 (Other: ANSM)
Record Dates: First submitted 2022-10-20; First posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Aging
MeSH Terms: interventions — Injections

STUDY DESIGN:
Intervention Model Description: 145 subjects divided into 2 groups (Randomization 3:1 for the face):
  • 107 subjects in treatment group on the face. Among these patients, N=55 were injected on the neck and N=49 on the décolleté.
  38 patients were included in the control group. Among these patients, all were studied on the neck and N=34 were studied on the décolleté
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Face and neck injection (Experimental): NCTF135HA intradermal injection on face and neck. 3 injections spaced out by two weeks; injection points are spaced every 1-1.5 cm with a quantity of 0.05 ml on each point.
  Application of Hydra Filler cream twice daily on the face and neck.
  Interventions: Device: injection
- Face and upper chest/décolleté injection (Experimental): NCTF135HA intradermal injection on face and décolleté. 3 injections spaced out by two weeks; injection points are spaced every 1-1.5 cm with a quantity of 0.05 ml on each point.
  Application of Hydra Filler cream twice daily on the face and décolleté.
  Interventions: Device: injection
- Face and neck controle (Active Comparator): Application of Hydra Filler cream twice daily on the face and neck.
  Interventions: Other: Cream application
- Face and upper chest/décolleté controle (Active Comparator): Application of Hydra Filler cream twice daily on the face and décolleté.
  Interventions: Other: Cream application

INTERVENTIONS:
Device: injection — Intradermal injection on the face and neck/or décolleté by the NCTF135 HA
  Arms: Face and neck injection; Face and upper chest/décolleté injection
Other: Cream application — Application of hydra filler cream on the face and neck/or décolleté
  Arms: Face and neck controle; Face and upper chest/décolleté controle

SUMMARY:
The NCTF135HA medical device from Laboratoires FILL-MED by FILORGA Company is an injectable solution for the treatment of wrinkles and biorevitalization of injected mature skin using a multi-injection technique with CE marking. It is a viscoelastic injectable solution of 1% hyaluronic acid (10mg/ml), non-crosslinked of non-animal origin, obtained by biofermentation, resorbable, opalescent, sterile and apyrogenic. NCTF135HA is an anti-aging viscoelastic solution for the revitalization and intense hydration of tired or dull skin, the treatment of wrinkles and the redensification of mature or sagging skin. This hyaluronic acid solution is intended to be injected into the superficial dermis to compensate for the loss of moisture. Given the expected impact of the injection procedure of the biorevitalization solution on wrinkles, the primary endpoint was chosen to evaluate the effectiveness of the treatment on wrinkles.

DETAILED DESCRIPTION:
Aging is a complex phenomenon that includes many structural changes over time. At the level of the face, the ageing of the superficial plane (skin) and that of the support structures (fat, muscles and bones) are distinguished. On the skin, there is a reduction in cell renewal, dehydration, loss of radiance, elasticity, firmness and the appearance of fine lines and wrinkles. The NCTF135HA medical device from Laboratoires FILL-MED by FILORGA Company is an injectable solution for the treatment of wrinkles and biorevitalization of injected mature skin using a multi-injection technique with CE marking. It is a viscoelastic injectable solution of 1% hyaluronic acid (10mg/ml), non-crosslinked of non-animal origin, obtained by biofermentation, resorbable, opalescent, sterile and apyrogenic. NCTF135HA is an anti-aging viscoelastic solution for the revitalization and intense hydration of tired or dull skin, the treatment of wrinkles and the redensification of mature or sagging skin. This hyaluronic acid solution is intended to be injected into the superficial dermis to compensate for the loss of moisture. Given the nature of the process under study, it is difficult to propose as a control a solution that includes only saline as an injection product. Indeed, the subject would suffer harm related to injections without a priori benefiting from them. In addition, a DM injected using a multi-injection technique is a whole combining micro-injections by themselves and the products injected. Therefore, it is proposed to use as a control group subjects who will be evaluated in a similar way to those treated by injections of the biorevitalization solution but whose only cosmetic care will consist of the application of a moisturizing cream. This cream, used daily, will also be applied by the subjects in the injection group Given the expected impact of the injection procedure of the biorevitalization solution on wrinkles, the primary endpoint was chosen to evaluate the effectiveness of the treatment on wrinkles. For the face, this criterion will be the evolution of the average volume of crow's feet wrinkles (depth and surface). It will be measured centrally by a validated 3D imaging technique. For the neck and décolleté areas that will also be studied, this assessment will be replaced by clinical scoring using photographic scales developed specifically for these areas (the typology of this type of wrinkle does not lend itself to conventional 3D analysis measurements). This evaluation will be completed by a series of other dermatological explorations, also non-invasive: clinical scoring, measurement of skin hydration, elasticity, photographic evaluation of skin ageing and measurement of dermal density by high frequency ultrasound

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥19 years old;
* Subject who has signed a written informed consent;
* Subject with a Fitzpatrick phototype of I, II, III or IV
* Subject with a grade of photoaging of 2 or 3 on a scale of Glogau
* Subject having a wrinkle score according to Lemperle scale of 2, 3 or 4 at the level of periorbital lines
* Subject having at least:

  * a Grade 1, 2, 3 or 4 on Bazin Neck Wrinkle Scale (at least N=30 subject for the control group)
  * or a Grade 2, 3 or 4 on Landau Décolleté Wrinkle Scale (at least N=30 subject for the control group)
* Subject registered in social security system or other health insurance regimen
* Subject accepting not to expose Him/herself to the sun or ultraviolet (UV) during the entire duration of the study.
* Female subject accepting to take a pregnancy test.

Exclusion Criteria:

* Subject involved in any other clinical study evaluating drugs or medical devices or subjects in exclusion periods of another clinical study.
* Subject deprived of freedom by an administrative or legal decision
* Unable to follow protocol requirements.
* Subject who has received indemnification of 4500 € during the 12 previous months for his/her participation in clinical trials (including participation in this study).
* Subject having benefited from injection/facial implantation of any non-absorbable filling agent at any time of his/her life.
* Subject having already had laser sessions for skin rejuvenation or a laser facelift in the previous year or a facelift by surgery in the 2 years prior to the study.
* Subject with a history of fillers injections (hyaluronic acid type) in the last year or botulinum toxin in the last 6 months or the injectable implants (semi-permanent fillers) in the last two years.
* Subject with a skin support device (wire mesh, gold wire, liquid silicone or other particulate material) at the study zones.
* Subject having done a moderate to deep peeling or non-invasive rejuvenation techniques such as radiofrequency, ultrasound and lasers in the last 6 months.
* Subject with a history of multiple severe allergies or anaphylactic shock.
* Subject with a known hypersensitivity to hyaluronic acid, or other components of the NCTF 135HA solution.
* Subject with known intolerance/hypersensitivity to any cosmetic topical products, hyaluronic acid and/or other components of Hydra-Filler ® FILORGA Moisturizing Cream.
* Subject with a known hypersensitivity to chlorhexidine.
* Subject with a known hypersensitivity to lidocaine or to local amide-type anesthetics
* Prone to developing inflammatory skin conditions or hypertrophic scarring according to investigator judgement.
* Subject with a history of streptococcal diseases (angina recurrent, rheumatic fever).
* Subject under concomitant treatment (or not stopped for at least 3 months) by oral or injectable corticosteroid (inhaled corticosteroids are allowed as well as a topical corticotherapy not involving the study zones).
* Subject under concomitant treatment (or not stopped for at least 1 year) by immunosuppressive or chemotherapy treatments.
* Subject with a history of less than one year of radiation therapy at the head and neck.
* Subject with an associated antecedent or pathology of autoimmune or connective tissue disease.
* Subject presenting a skin pathology, an acute inflammatory reaction or a bacterial or viral infection on the study zones or within the 6 weeks after the end of such an episode.
* Subject having taken aspirin or anticoagulants, at regular doses, in the last 15 days preceding the act.
* Subject that has been exposed to sun or UV in the last 15 days.
* Subject with a dermatological condition or inflammation at the treatment zone or near to this area (according to the investigator's judgment).
* Pregnant or lactating woman (Before every injection, a urinary pregnancy test will be performed).
* Subject having epilepsy uncontrolled by treatment.
* Subject presenting a general pathology, skin pathology, dermatosis, systemic, chronic or acute disease and/or topical or general treatment that in the opinion of the investigator may interfere with the treatment or compromise the participation of the subject in the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-11-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline of the mean volume of crow's feet wrinkles for the face at Day 75 | Day 75 (75 days after the injection
  Change from Baseline of the mean volume of crow's feet wrinkles for the face at Day 75 e (depth and surface) in mm^3 measured by LifeViz 3D micro® of injected group compared to control group

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Jean-Jacques DEUTSCH, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fanian F, Deutsch JJ, Bousquet MT, Boisnic S, Andre P, Catoni I, Beilin G, Lemmel C, Taieb M, Gomel-Toledano M, Issa H, Garcia P. A hyaluronic acid-based micro-filler improves superficial wrinkles and skin quality: a randomized prospective controlled multicenter study. J Dermatolog Treat. 2023 Dec;34(1):2216323. doi: 10.1080/09546634.2023.2216323. Epub 2023 Aug 14. PMID 37577796